CLINICAL TRIAL: NCT06117800
Title: Effect of Evidence Based Teamwork System on Patient Safety Culture Among Newly Graduate Nurses at Main Mansoura University Hospital
Brief Title: Effect of Evidence Based Teamwork System on Patient Safety Culture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asmaa Elwan Mohammed Hassan (Other)
Responsible Party: Sponsor-Investigator, Asmaa Elwan Mohammed Hassan, Assistant lecturer of Nursing Administration Faculty of Nursing, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TeamSTEPPS
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Team STEPPS and Patient Safety Culture (Experimental): TeamSTEPPS®) is an evidence-based framework that has been used in interprofessional education programs to develop and train newly graduate nurses to deal with difficult clinical situations. Patient safety culture means preventing unintended incidents or accidents that may happen in a certain period in serving health care to patients
  Interventions: Other: TeamSTEPPS

INTERVENTIONS:
Other: TeamSTEPPS — Team Tools and Strategies to Enhance Performance and Patient Safety (TeamSTEPPS®) is an evidence-based framework that has been used in interprofessional education programs to develop and train newly graduate nurses to deal with difficult clinical situations.

SUMMARY:
This study aims to evaluate the effect of evidence-based teamwork system on patient safety culture among newly graduate nurses at Main Mansoura University Hospital

DETAILED DESCRIPTION:
Developing a patient safety culture was one of the recommendations made by the Institute of Medicine to assist hospitals in improving patient safety and crucial for healthcare quality. Newly graduated nurses with lower levels of work experience, education, and work as part of a team in the healthcare setting are needed to develop communication and teamwork skill to improve patient safety culture . Ineffective communication and teamwork skill among newly graduated nurses are associated with negative patient safety culture outcomes, such as increased error rates, increased length of hospital stay, medication errors, pressure ulcers, and death. The implementation of modified TeamSTEPPS is highly expected to promote better interprofessional communication and teamwork skill between newly graduate nurses as well as improve patient safety culture. So that, this study aims to evaluate the effect of evidence-based teamwork system on patient safety culture among newly graduate nurses at Main Mansoura University Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. All full-time and part-time newly graduated nurses in all departments at Main Mansoura University Hospital within the last two years,
2. Who provide direct patient care
3. Willing to participate in the study.

Exclusion Criteria:

1. All newly graduated nurses who graduated more than two years
2. Who do not provide direct patient care were excluded from the study.
3. All newly graduated nurses through an outside registry or contract through a third party, on a per diem basis
4. Who floated to the intervention unit from another unit were excluded from the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
The newly graduated nurses' perceptions about patient safety culture as assessed by (HSPSC)Tool | from start to finish, up to three month
  The Hospital Survey on Patient Safety Culture (HSPSC) Tool is survey that designed by The Agency for Healthcare Research and Quality specifically for hospital staff and used to determine the newly graduated nurses' perceptions about the culture of patient safety before and after implementing the program.

SECONDARY OUTCOMES:
Improve the patient safety culture for newly graduated nurses through the implementation of (TeamSTEPPS) training program and assessed by (T-TPQ) survey tool. | from start to finish, up to three month
  The Team STEPPS Teamwork Perceptions Questionnaire (T-TPQ) Survey is tool that designed by The Agency for Healthcare Research and Quality and used to evaluate the effectiveness TeamSTEPPS® training on patient safety culture among newly graduated nurses before and after implementing the program.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Elwan Mohammed Hassan, Doctorate, Principal Investigator — Faculty of Nursing -Mansoura University
Locations (1):
- Faculty of Nursing -Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Gaston T, Short N, Ralyea C, Casterline G. Promoting Patient Safety: Results of a TeamSTEPPS(R) Initiative. J Nurs Adm. 2016 Apr;46(4):201-7. doi: 10.1097/NNA.0000000000000333. PMID 27011154
- [Result] Rosen MA, DiazGranados D, Dietz AS, Benishek LE, Thompson D, Pronovost PJ, Weaver SJ. Teamwork in healthcare: Key discoveries enabling safer, high-quality care. Am Psychol. 2018 May-Jun;73(4):433-450. doi: 10.1037/amp0000298. PMID 29792459
- [Result] Sweigart LI, Umoren RA, Scott PJ, Carlton KH, Jones JA, Truman B, Gossett EJ. Virtual TeamSTEPPS((R)) Simulations Produce Teamwork Attitude Changes Among Health Professions Students. J Nurs Educ. 2016 Jan;55(1):31-5. doi: 10.3928/01484834-20151214-08. PMID 26812380
- See also: The effects of simulation based TeamSTEPPS interprofessional communication and teamwork training on patient and provider outcomes (Doctoral dissertation, UCLA). — http://escholarship.org/uc/item/6xz705jf